CLINICAL TRIAL: NCT03671746
Title: Inflammatory Response to Trauma - Does Early Cytokine Modulation Improve Patient Outcome
Brief Title: Inflammatory Markers in Trauma Patient Outcomes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arun Aneja (Other)
Responsible Party: Sponsor-Investigator, Arun Aneja, Assistant Professor of Orthopaedic Surgery Traumatology Division, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 43611
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Polytrauma
Keywords: Inflammatory cytokine; inflammation; trauma; opioid
MeSH Terms: conditions — Multiple Trauma; Inflammation; Wounds and Injuries | interventions — Ketorolac; Ketorolac Tromethamine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Compare the effectiveness of a NSAID to placebo in acute trauma setting.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participant medical team will be blinded to the treatment or placebo intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care without NSAID (Placebo Comparator): Polytrauma participants will receive standard of care in addition to saline solution according to standard Advanced Trauma Life Support (ATLS) and standard ICU routine medical care.
  Interventions: Drug: Saline Solution
- Standard of Care with NSAID (Experimental): Participants in the group will receive Ketorolac in addition to standard of care for the standard Advanced Trauma Life Support (ATLS) and standard ICU routine medical care.
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — Participants will receive Ketorolac at 15 mg IV every 6 hours for their first 5 days of hospitalization
  Other Names: Toradol
  Arms: Standard of Care with NSAID
Drug: Saline Solution — Participants will receive 1 ml of saline solution IV every 6 hours for their first 5 days of hospitalization
  Other Names: Normal Saline
  Arms: Standard of Care without NSAID

SUMMARY:
It is unknown whether early modulation of inflammatory cytokines is associated with improved patient outcomes, reduced narcotic requirements in orthopaedic patient population, and improved patient subjective pain after hospital discharge. Preliminary animal and clinical studies have shown correlation between elevated blood cytokine concentrations during the acute phase of trauma and the development of post-traumatic complications. Early administration of nonsteroidal anti-inflammatory drug (NSAID) in animals significantly reduced inflammatory profiles, improved pulmonary edema, and enhanced arteriole vasoconstriction in response to hemorrhage. The ability to modify post-traumatic physiologic response via short-term administration of a non-steroidal anti-inflammatory drug (NSAID) may lead to improved patient outcome. In addition, given the current landscape for opioid epidemic in the United States, alternative non-opioid pain management during acute trauma has the potential to reduce opioid consumption and represents a pivotal component of multimodal analgesia strategy.

By doing this study, the investigators hope to learn how to provide the best care for all patients in the state of Kentucky. Patient participation in this research will last about 1 year.

DETAILED DESCRIPTION:
Accidental trauma is the 4th leading cause of death in the United States, and it is associated with a complex inflammatory response. This response is associated with post-traumatic complications such as; multi-organ dysfunction syndrome (MODS), bacterial pneumonia, acute respiratory distress syndrome (ARDS), systemic inflammatory response syndrome (SIRS), and post-traumatic pain (PTP). It is unknown whether early modulation of inflammatory cytokines is associated with improved patient outcomes, reduced narcotic requirements, and improved patient subjective pain after hospital discharge.

Preliminary data has shown: (1) elevated blood cytokine concentrations during the acute phase of trauma are correlated with the development of fatal post-traumatic complications, (2) that early administration of a non-steroidal anti-inflammatory drug (NSAID) resulted in decreased blood serum levels of interleukin (IL-6), Prostaglandin E2 (PGE2), improved pulmonary edema, and enhanced arterioles ability to vasoconstrict in response to hemorrhage in animal models, and (3) that the addition of the internal physiologic parameters (inflammatory cytokines) to New Injury Severity Score (NISS - a marker of the external anatomical insult) significantly improves the ability to predict hospital length of stay of trauma patients when compared to NISS alone. The investigator's group is the first to use an integrative approach that combines the external anatomic injury data with the internal physiologic response for accurate prediction of a patient's clinical outcome. Therefore, if the investigators apply this same mindset to treatment, the investigators can improve the trauma patients' care by addressing both parameters as opposed to solely focusing on the external injury as done in the past. The ability to modify post-traumatic physiologic response via short-term administration of an NSAID may lead to improved patient outcomes.

Over the last decade, clinicians have remained puzzled over the safety of NSAID administration after fracture in terms of bone union. In addition, given the current landscape for the opioid epidemic in the United States, alternative non-opioid pain management during acute trauma has the potential to reduce opioid consumption and represents a pivotal component of multimodal analgesia strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 to 75
* New Injury Severity Score (NISS) > 9, with musculoskeletal injury requiring surgical treatment

Exclusion Criteria:

* Patient age < 18 or > 75
* Patients who presented more than 24 hours after time of injury
* Patients with contraindications to NSAID therapy (i.e., patients with active hemorrhage, received blood products, traumatic brain injury (TBI), active gastrointestinal bleeding or ulceration, NSAID allergy, thromboembolism, or coagulopathy)
* Patients with pre-existing inflammatory condition (e.g., inflammatory arthropathy or bowel disease)
* Patients with preexisting immunocompromised/immunosuppressed condition or acquired immunodeficiency syndrome (AIDS)
* Patients with pre-existing comorbidities (e.g., coronary artery disease, myocardial infarction, chronic organ failure, chronic obstructive pulmonary disease, emphysema, asthma, etc.)
* Patients with chronic use of steroids, immuno-modulating drugs, or history of organ transplantation
* Patients receiving chronic opioid therapy or treatment for opioid use disorder
* Patients who are pregnant
* Patients with thermal injury

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arun Aneja, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braden JB, Fan MY, Edlund MJ, Martin BC, DeVries A, Sullivan MD. Trends in use of opioids by noncancer pain type 2000-2005 among Arkansas Medicaid and HealthCore enrollees: results from the TROUP study. J Pain. 2008 Nov;9(11):1026-35. doi: 10.1016/j.jpain.2008.06.002. Epub 2008 Jul 26. PMID 18676205
- [Background] Lawal OD, Gold J, Murthy A, Ruchi R, Bavry E, Hume AL, Lewkowitz AK, Brothers T, Wen X. Rate and Risk Factors Associated With Prolonged Opioid Use After Surgery: A Systematic Review and Meta-analysis. JAMA Netw Open. 2020 Jun 1;3(6):e207367. doi: 10.1001/jamanetworkopen.2020.7367. PMID 32584407
- [Background] Mohamadi A, Chan JJ, Lian J, Wright CL, Marin AM, Rodriguez EK, von Keudell A, Nazarian A. Risk Factors and Pooled Rate of Prolonged Opioid Use Following Trauma or Surgery: A Systematic Review and Meta-(Regression) Analysis. J Bone Joint Surg Am. 2018 Aug 1;100(15):1332-1340. doi: 10.2106/JBJS.17.01239. PMID 30063596
- [Background] Bosse MJ, MacKenzie EJ, Kellam JF, Burgess AR, Webb LX, Swiontkowski MF, Sanders RW, Jones AL, McAndrew MP, Patterson BM, McCarthy ML, Travison TG, Castillo RC. An analysis of outcomes of reconstruction or amputation after leg-threatening injuries. N Engl J Med. 2002 Dec 12;347(24):1924-31. doi: 10.1056/NEJMoa012604. PMID 12477942
- [Background] Castillo RC, MacKenzie EJ, Webb LX, Bosse MJ, Avery J; LEAP Study Group. Use and perceived need of physical therapy following severe lower-extremity trauma. Arch Phys Med Rehabil. 2005 Sep;86(9):1722-8. doi: 10.1016/j.apmr.2005.03.005. PMID 16181933
- [Background] O'Toole RV, Castillo RC, Pollak AN, MacKenzie EJ, Bosse MJ; LEAP Study Group. Determinants of patient satisfaction after severe lower-extremity injuries. J Bone Joint Surg Am. 2008 Jun;90(6):1206-11. doi: 10.2106/JBJS.G.00492. PMID 18519312
- [Background] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Background] Sherwood GD, McNeill JA, Starck PL, Disnard G. Changing acute pain management outcomes in surgical patients. AORN J. 2003 Feb;77(2):374, 377-80, 384-90 passim. doi: 10.1016/s0001-2092(06)61206-4. PMID 12619852
- [Background] Hsu JR, Mir H, Wally MK, Seymour RB; Orthopaedic Trauma Association Musculoskeletal Pain Task Force. Clinical Practice Guidelines for Pain Management in Acute Musculoskeletal Injury. J Orthop Trauma. 2019 May;33(5):e158-e182. doi: 10.1097/BOT.0000000000001430. PMID 30681429
- [Background] Oyler DR, Slade E, Slavova S, Matuszewski PE, Lei F, Herndon B, Johnson S, Moghadamian ES. Effect of a Multimodal Analgesic Protocol on Short-Term and Long-Term Opioid Use After Orthopaedic Trauma. J Orthop Trauma. 2022 Aug 1;36(8):326-331. doi: 10.1097/BOT.0000000000002346. Epub 2022 Jan 6. PMID 34999625
- [Background] Mir HR, Miller AN, Obremskey WT, Jahangir AA, Hsu JR. Confronting the Opioid Crisis: Practical Pain Management and Strategies: AOA 2018 Critical Issues Symposium. J Bone Joint Surg Am. 2019 Dec 4;101(23):e126. doi: 10.2106/JBJS.19.00285. PMID 31800430
- [Background] Castillo RC, Raja SN, Frey KP, Vallier HA, Tornetta P 3rd, Jaeblon T, Goff BJ, Gottschalk A, Scharfstein DO, O'Toole RV; METRC. Improving Pain Management and Long-Term Outcomes Following High-Energy Orthopaedic Trauma (Pain Study). J Orthop Trauma. 2017 Apr;31 Suppl 1:S71-S77. doi: 10.1097/BOT.0000000000000793. PMID 28323806
- [Background] Marquez-Lara A, Hutchinson ID, Nunez F Jr, Smith TL, Miller AN. Nonsteroidal Anti-Inflammatory Drugs and Bone-Healing: A Systematic Review of Research Quality. JBJS Rev. 2016 Mar 15;4(3):e4. doi: 10.2106/JBJS.RVW.O.00055. PMID 27500434
- [Background] Cepeda MS, Carr DB, Miranda N, Diaz A, Silva C, Morales O. Comparison of morphine, ketorolac, and their combination for postoperative pain: results from a large, randomized, double-blind trial. Anesthesiology. 2005 Dec;103(6):1225-32. doi: 10.1097/00000542-200512000-00018. PMID 16306736
- [Background] McDonald EL, Daniel JN, Rogero RG, Shakked RJ, Nicholson K, Pedowitz DI, Raikin SM, Bilolikar V, Winters BS. How Does Perioperative Ketorolac Affect Opioid Consumption and Pain Management After Ankle Fracture Surgery? Clin Orthop Relat Res. 2020 Jan;478(1):144-151. doi: 10.1097/CORR.0000000000000978. PMID 31567579
- [Background] Vadivelu N, Gowda AM, Urman RD, Jolly S, Kodumudi V, Maria M, Taylor R Jr, Pergolizzi JV Jr. Ketorolac tromethamine - routes and clinical implications. Pain Pract. 2015 Feb;15(2):175-93. doi: 10.1111/papr.12198. Epub 2014 Apr 16. PMID 24738596
- [Background] Brown CR, Mazzulla JP, Mok MS, Nussdorf RT, Rubin PD, Schwesinger WH. Comparison of repeat doses of intramuscular ketorolac tromethamine and morphine sulfate for analgesia after major surgery. Pharmacotherapy. 1990;10(6 ( Pt 2)):45S-50S. PMID 2082313
- [Background] Camu F, Van Overberge L, Bullingham R, Lloyd J. Hemodynamic effects of two intravenous doses of ketorolac tromethamine compared with morphine. Pharmacotherapy. 1990;10(6 ( Pt 2)):122S-126S. PMID 2082308
- [Background] De Oliveira GS Jr, Agarwal D, Benzon HT. Perioperative single dose ketorolac to prevent postoperative pain: a meta-analysis of randomized trials. Anesth Analg. 2012 Feb;114(2):424-33. doi: 10.1213/ANE.0b013e3182334d68. Epub 2011 Sep 29. PMID 21965355
- [Background] Jelinek GA. Ketorolac versus morphine for severe pain. Ketorolac is more effective, cheaper, and has fewer side effects. BMJ. 2000 Nov 18;321(7271):1236-7. doi: 10.1136/bmj.321.7271.1236. No abstract available. PMID 11082068
- [Background] Gobble RM, Hoang HLT, Kachniarz B, Orgill DP. Ketorolac does not increase perioperative bleeding: a meta-analysis of randomized controlled trials. Plast Reconstr Surg. 2014 Mar;133(3):741-755. doi: 10.1097/01.prs.0000438459.60474.b5. PMID 24572864
- [Background] Irizarry E, Restivo A, Salama M, Davitt M, Feliciano C, Cortijo-Brown A, Friedman BW. A randomized controlled trial of ibuprofen versus ketorolac versus diclofenac for acute, nonradicular low back pain. Acad Emerg Med. 2021 Nov;28(11):1228-1235. doi: 10.1111/acem.14321. Epub 2021 Jun 30. PMID 34133820
- [Background] Motov S, Yasavolian M, Likourezos A, Pushkar I, Hossain R, Drapkin J, Cohen V, Filk N, Smith A, Huang F, Rockoff B, Homel P, Fromm C. Comparison of Intravenous Ketorolac at Three Single-Dose Regimens for Treating Acute Pain in the Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2017 Aug;70(2):177-184. doi: 10.1016/j.annemergmed.2016.10.014. Epub 2016 Dec 16. PMID 27993418
- [Background] Gillis JC, Brogden RN. Ketorolac. A reappraisal of its pharmacodynamic and pharmacokinetic properties and therapeutic use in pain management. Drugs. 1997 Jan;53(1):139-88. doi: 10.2165/00003495-199753010-00012. PMID 9010653
- [Background] Kinsella J, Moffat AC, Patrick JA, Prentice JW, McArdle CS, Kenny GN. Ketorolac trometamol for postoperative analgesia after orthopaedic surgery. Br J Anaesth. 1992 Jul;69(1):19-22. doi: 10.1093/bja/69.1.19. PMID 1303630
- [Background] Reinhart DI. Minimising the adverse effects of ketorolac. Drug Saf. 2000 Jun;22(6):487-97. doi: 10.2165/00002018-200022060-00007. PMID 10877042
- [Background] Lavoie A, Moore L, LeSage N, Liberman M, Sampalis JS. The New Injury Severity Score: a more accurate predictor of in-hospital mortality than the Injury Severity Score. J Trauma. 2004 Jun;56(6):1312-20. doi: 10.1097/01.ta.0000075342.36072.ef. PMID 15211142
- [Background] Lavoie A, Moore L, LeSage N, Liberman M, Sampalis JS. The Injury Severity Score or the New Injury Severity Score for predicting intensive care unit admission and hospital length of stay? Injury. 2005 Apr;36(4):477-83. doi: 10.1016/j.injury.2004.09.039. Epub 2005 Jan 22. PMID 15755427
- [Background] Weisz RD, Fokin AA, Lerner V, Flynt A, Macias-Perez I, Pavliv L, Crawford M, Puente I. Intravenous Ibuprofen Reduces Opioid Consumption During the Initial 48 Hours After Injury in Orthopedic Trauma Patients. J Orthop Trauma. 2020 Jul;34(7):341-347. doi: 10.1097/BOT.0000000000001733. PMID 31929374
- [Background] Singla N, Rock A, Pavliv L. A multi-center, randomized, double-blind placebo-controlled trial of intravenous-ibuprofen (IV-ibuprofen) for treatment of pain in post-operative orthopedic adult patients. Pain Med. 2010 Aug;11(8):1284-93. doi: 10.1111/j.1526-4637.2010.00896.x. Epub 2010 Jun 30. PMID 20609131
- [Background] Southworth S, Peters J, Rock A, Pavliv L. A multicenter, randomized, double-blind, placebo-controlled trial of intravenous ibuprofen 400 and 800 mg every 6 hours in the management of postoperative pain. Clin Ther. 2009 Sep;31(9):1922-35. doi: 10.1016/j.clinthera.2009.08.026. PMID 19843482
- [Background] Zhou HS, Li TT, Pi Y, Wang TH, Liu F, Xiong LL. Analgesic Efficacy of Intravenous Ibuprofen in the Treatment of Postoperative Acute Pain: A Phase III Multicenter Randomized Placebo-ControlledDouble-Blind Clinical Trial. Pain Res Manag. 2023 Mar 7;2023:7768704. doi: 10.1155/2023/7768704. eCollection 2023. PMID 36926379
- [Background] Eberson CP, Pacicca DM, Ehrlich MG. The role of ketorolac in decreasing length of stay and narcotic complications in the postoperative pediatric orthopaedic patient. J Pediatr Orthop. 1999 Sep-Oct;19(5):688-92. PMID 10488877
- [Background] Ellis TA 2nd, Hammoud H, Dela Merced P, Nooli NP, Ghoddoussi F, Kong J, Krishnan SH. Multimodal Clinical Pathway With Adductor Canal Block Decreases Hospital Length of Stay, Improves Pain Control, and Reduces Opioid Consumption in Total Knee Arthroplasty Patients: A Retrospective Review. J Arthroplasty. 2018 Aug;33(8):2440-2448. doi: 10.1016/j.arth.2018.03.053. Epub 2018 Mar 27. PMID 29691180
- [Background] Johnson P, Hustedt J, Matiski T, Childers R, Lederman E. Improvement in Postoperative Pain Control and Length of Stay With Peripheral Nerve Block Prior to Distal Radius Repair. Orthopedics. 2020 Nov 1;43(6):e549-e552. doi: 10.3928/01477447-20200721-14. Epub 2020 Aug 6. PMID 32745216
- [Background] Walker CT, Gullotti DM, Prendergast V, Radosevich J, Grimm D, Cole TS, Godzik J, Patel AA, Whiting AC, Little A, Uribe JS, Kakarla UK, Turner JD. Implementation of a Standardized Multimodal Postoperative Analgesia Protocol Improves Pain Control, Reduces Opioid Consumption, and Shortens Length of Hospital Stay After Posterior Lumbar Spinal Fusion. Neurosurgery. 2020 Jul 1;87(1):130-136. doi: 10.1093/neuros/nyz312. PMID 31414128
- [Background] Archer KR, Castillo RC, Wegener ST, Abraham CM, Obremskey WT. Pain and satisfaction in hospitalized trauma patients: the importance of self-efficacy and psychological distress. J Trauma Acute Care Surg. 2012 Apr;72(4):1068-77. doi: 10.1097/TA.0b013e3182452df5. PMID 22491629
- [Background] Bot AG, Bekkers S, Arnstein PM, Smith RM, Ring D. Opioid use after fracture surgery correlates with pain intensity and satisfaction with pain relief. Clin Orthop Relat Res. 2014 Aug;472(8):2542-9. doi: 10.1007/s11999-014-3660-4. Epub 2014 Apr 29. PMID 24777731
- [Background] Nota SP, Spit SA, Voskuyl T, Bot AG, Hageman MG, Ring D. Opioid Use, Satisfaction, and Pain Intensity After Orthopedic Surgery. Psychosomatics. 2015 Sep-Oct;56(5):479-85. doi: 10.1016/j.psym.2014.09.003. Epub 2014 Sep 6. PMID 25624183
- [Background] Shah A, Hayes CJ, Martin BC. Characteristics of Initial Prescription Episodes and Likelihood of Long-Term Opioid Use - United States, 2006-2015. MMWR Morb Mortal Wkly Rep. 2017 Mar 17;66(10):265-269. doi: 10.15585/mmwr.mm6610a1. PMID 28301454
- [Background] Morris BJ, Mir HR. The opioid epidemic: impact on orthopaedic surgery. J Am Acad Orthop Surg. 2015 May;23(5):267-71. doi: 10.5435/JAAOS-D-14-00163. PMID 25911660
- [Background] Rodriguez-Buitrago A, Attum B, Enata N, Evans A, Okwumabua E, Gajari V, Obremskey WT, Jahangir A. Opiate Prescribing Practices After Common Isolated Lower Extremity Injuries. J Orthop Trauma. 2019 Mar;33(3):e93-e99. doi: 10.1097/BOT.0000000000001375. PMID 30779727
- [Background] Castillo RC, MacKenzie EJ, Wegener ST, Bosse MJ; LEAP Study Group. Prevalence of chronic pain seven years following limb threatening lower extremity trauma. Pain. 2006 Oct;124(3):321-329. doi: 10.1016/j.pain.2006.04.020. Epub 2006 Jun 15. PMID 16781066
- [Background] von Oelreich E, Eriksson M, Brattstrom O, Sjolund KF, Discacciati A, Larsson E, Oldner A. Risk factors and outcomes of chronic opioid use following trauma. Br J Surg. 2020 Mar;107(4):413-421. doi: 10.1002/bjs.11507. Epub 2020 Feb 7. PMID 32031251
- [Background] Norman SB, Stein MB, Dimsdale JE, Hoyt DB. Pain in the aftermath of trauma is a risk factor for post-traumatic stress disorder. Psychol Med. 2008 Apr;38(4):533-42. doi: 10.1017/S0033291707001389. Epub 2007 Sep 10. PMID 17825121
- [Background] Oostinga D, Steverink JG, van Wijck AJM, Verlaan JJ. An understanding of bone pain: A narrative review. Bone. 2020 May;134:115272. doi: 10.1016/j.bone.2020.115272. Epub 2020 Feb 13. PMID 32062002
- [Background] Martin BC, Fan MY, Edlund MJ, Devries A, Braden JB, Sullivan MD. Long-term chronic opioid therapy discontinuation rates from the TROUP study. J Gen Intern Med. 2011 Dec;26(12):1450-7. doi: 10.1007/s11606-011-1771-0. Epub 2011 Jul 13. PMID 21751058
- [Background] Van Zee A. The promotion and marketing of oxycontin: commercial triumph, public health tragedy. Am J Public Health. 2009 Feb;99(2):221-7. doi: 10.2105/AJPH.2007.131714. Epub 2008 Sep 17. PMID 18799767
- [Background] White PF. The changing role of non-opioid analgesic techniques in the management of postoperative pain. Anesth Analg. 2005 Nov;101(5 Suppl):S5-S22. doi: 10.1213/01.ANE.0000177099.28914.A7. PMID 16334489
- [Background] Choban PS, Weireter LJ Jr, Maynes C. Obesity and increased mortality in blunt trauma. J Trauma. 1991 Sep;31(9):1253-7. doi: 10.1097/00005373-199109000-00009. PMID 1920556
- [Background] Roberts CS, Pape HC, Jones AL, Malkani AL, Rodriguez JL, Giannoudis PV. Damage control orthopaedics: evolving concepts in the treatment of patients who have sustained orthopaedic trauma. Instr Course Lect. 2005;54:447-62. PMID 15948472
- [Background] DeLong WG Jr, Born CT. Cytokines in patients with polytrauma. Clin Orthop Relat Res. 2004 May;(422):57-65. doi: 10.1097/01.blo.0000130840.64528.1e. PMID 15187834
- [Background] McKinley TO, Gaski GE, Vodovotz Y, Corona BT, Billiar TR. Diagnosis and Management of Polytraumatized Patients With Severe Extremity Trauma. J Orthop Trauma. 2018 Mar;32 Suppl 1:S1-S6. doi: 10.1097/BOT.0000000000001114. PMID 29461394
- [Background] Brochner AC, Toft P. Pathophysiology of the systemic inflammatory response after major accidental trauma. Scand J Trauma Resusc Emerg Med. 2009 Sep 15;17:43. doi: 10.1186/1757-7241-17-43. PMID 19754938
- [Background] Tsirigotis P, Chondropoulos S, Gkirkas K, Meletiadis J, Dimopoulou I. Balanced control of both hyper and hypo-inflammatory phases as a new treatment paradigm in sepsis. J Thorac Dis. 2016 May;8(5):E312-6. doi: 10.21037/jtd.2016.03.47. PMID 27162689
- [Background] Cuschieri J, Bulger E, Schaeffer V, Sakr S, Nathens AB, Hennessy L, Minei J, Moore EE, O'Keefe G, Sperry J, Remick D, Tompkins R, Maier RV; Inflammation and the Host Response to Injury Collaborative Research Program. Early elevation in random plasma IL-6 after severe injury is associated with development of organ failure. Shock. 2010 Oct;34(4):346-51. doi: 10.1097/SHK.0b013e3181d8e687. PMID 20844410
- [Background] Frink M, Hsieh YC, Hsieh CH, Pape HC, Choudhry MA, Schwacha MG, Chaudry IH. Keratinocyte-derived chemokine plays a critical role in the induction of systemic inflammation and tissue damage after trauma-hemorrhage. Shock. 2007 Nov;28(5):576-81. doi: 10.1097/shk.0b013e31814b8e0d. PMID 18084824
- [Background] Giannoudis PV, Smith RM, Perry SL, Windsor AJ, Dickson RA, Bellamy MC. Immediate IL-10 expression following major orthopaedic trauma: relationship to anti-inflammatory response and subsequent development of sepsis. Intensive Care Med. 2000 Aug;26(8):1076-81. doi: 10.1007/s001340051320. PMID 11030163
- [Background] Hildebrand F, Giannoudis PV, van Griensven M, Chawda M, Pape HC. Pathophysiologic changes and effects of hypothermia on outcome in elective surgery and trauma patients. Am J Surg. 2004 Mar;187(3):363-71. doi: 10.1016/j.amjsurg.2003.12.016. PMID 15006564
- [Background] Pape HC, Schmidt RE, Rice J, van Griensven M, das Gupta R, Krettek C, Tscherne H. Biochemical changes after trauma and skeletal surgery of the lower extremity: quantification of the operative burden. Crit Care Med. 2000 Oct;28(10):3441-8. doi: 10.1097/00003246-200010000-00012. PMID 11057799
- [Background] Vanzant EL, Lopez CM, Ozrazgat-Baslanti T, Ungaro R, Davis R, Cuenca AG, Gentile LF, Nacionales DC, Cuenca AL, Bihorac A, Leeuwenburgh C, Lanz J, Baker HV, McKinley B, Moldawer LL, Moore FA, Efron PA. Persistent inflammation, immunosuppression, and catabolism syndrome after severe blunt trauma. J Trauma Acute Care Surg. 2014 Jan;76(1):21-9; discussion 29-30. doi: 10.1097/TA.0b013e3182ab1ab5. PMID 24368353
- [Background] Gaski GE, Metzger C, McCarroll T, Wessel R, Adler J, Cutshall A, Brown K, Vodovotz Y, Billiar TR, McKinley TO. Early Immunologic Response in Multiply Injured Patients With Orthopaedic Injuries Is Associated With Organ Dysfunction. J Orthop Trauma. 2019 May;33(5):220-228. doi: 10.1097/BOT.0000000000001437. PMID 31008819
- [Background] Stutz CM, O'Rear LD, O'Neill KR, Tamborski ME, Crosby CG, Devin CJ, Schoenecker JG. Coagulopathies in orthopaedics: links to inflammation and the potential of individualizing treatment strategies. J Orthop Trauma. 2013 Apr;27(4):236-41. doi: 10.1097/BOT.0b013e318269b782. PMID 22874115
- [Background] Adib-Conquy M, Cavaillon JM. Compensatory anti-inflammatory response syndrome. Thromb Haemost. 2009 Jan;101(1):36-47. PMID 19132187
- [Background] McKinley TO, Gaski GE, Zamora R, Shen L, Sun Q, Namas RA, Billiar TR, Vodovotz Y. Early dynamic orchestration of immunologic mediators identifies multiply injured patients who are tolerant or sensitive to hemorrhage. J Trauma Acute Care Surg. 2021 Mar 1;90(3):441-450. doi: 10.1097/TA.0000000000002998. PMID 33093290
- [Background] Waydhas C, Nast-Kolb D, Trupka A, Zettl R, Kick M, Wiesholler J, Schweiberer L, Jochum M. Posttraumatic inflammatory response, secondary operations, and late multiple organ failure. J Trauma. 1996 Apr;40(4):624-30; discussion 630-1. doi: 10.1097/00005373-199604000-00018. PMID 8614044
- [Background] Malik A, Kanneganti TD. Function and regulation of IL-1alpha in inflammatory diseases and cancer. Immunol Rev. 2018 Jan;281(1):124-137. doi: 10.1111/imr.12615. PMID 29247991
- [Background] Dinarello CA. Overview of the IL-1 family in innate inflammation and acquired immunity. Immunol Rev. 2018 Jan;281(1):8-27. doi: 10.1111/imr.12621. PMID 29247995
- [Background] Dinarello CA. Interleukin-1 in the pathogenesis and treatment of inflammatory diseases. Blood. 2011 Apr 7;117(14):3720-32. doi: 10.1182/blood-2010-07-273417. Epub 2011 Feb 8. PMID 21304099
- [Background] Aneja A, Landy DC, Mittwede PN, Albano AY, Teasdall RJ, Isla A, Kavolus M. Inflammatory cytokines associated with outcomes in orthopedic trauma patients independent of New Injury Severity score: A pilot prospective cohort study. J Orthop Res. 2022 Jul;40(7):1555-1562. doi: 10.1002/jor.25183. Epub 2021 Nov 2. PMID 34729810
- [Background] Berg DJ, Zhang J, Lauricella DM, Moore SA. Il-10 is a central regulator of cyclooxygenase-2 expression and prostaglandin production. J Immunol. 2001 Feb 15;166(4):2674-80. doi: 10.4049/jimmunol.166.4.2674. PMID 11160331
- [Background] Harizi H, Gualde N. Pivotal role of PGE2 and IL-10 in the cross-regulation of dendritic cell-derived inflammatory mediators. Cell Mol Immunol. 2006 Aug;3(4):271-7. PMID 16978535
- [Background] Chu CH, Chen SH, Wang Q, Langenbach R, Li H, Zeldin D, Chen SL, Wang S, Gao H, Lu RB, Hong JS. PGE2 Inhibits IL-10 Production via EP2-Mediated beta-Arrestin Signaling in Neuroinflammatory Condition. Mol Neurobiol. 2015 Aug;52(1):587-600. doi: 10.1007/s12035-014-8889-0. Epub 2014 Sep 14. PMID 25218510
- [Background] Spruijt NE, Visser T, Leenen LP. A systematic review of randomized controlled trials exploring the effect of immunomodulative interventions on infection, organ failure, and mortality in trauma patients. Crit Care. 2010;14(4):R150. doi: 10.1186/cc9218. Epub 2010 Aug 5. PMID 20687920
- [Background] Dionne RA, Khan AA, Gordon SM. Analgesia and COX-2 inhibition. Clin Exp Rheumatol. 2001 Nov-Dec;19(6 Suppl 25):S63-70. PMID 11695255
- [Background] Xiang L, Lu S, Fuller W, Aneja A, Russell GV, Jones LB, Hester R. Impaired blood pressure recovery to hemorrhage in obese Zucker rats with orthopedic trauma. Am J Physiol Heart Circ Physiol. 2012 Jan 1;302(1):H340-8. doi: 10.1152/ajpheart.00439.2011. Epub 2011 Oct 14. PMID 22003055
- [Background] Xiang L, Hester RL, Fuller WL, Sebai ME, Mittwede PN, Jones EK, Aneja A, Russell GV. Orthopedic trauma-induced pulmonary injury in the obese Zucker rat. Microcirculation. 2010 Nov;17(8):650-9. doi: 10.1111/j.1549-8719.2010.00061.x. PMID 21044219
- [Background] Peirce RJ, Fragen RJ, Pemberton DM. Intravenous ketorolac tromethamine versus morphine sulfate in the treatment of immediate postoperative pain. Pharmacotherapy. 1990;10(6 ( Pt 2)):111S-115S. PMID 2082306
- [Background] Lichtenstein DA, Meziere GA. Relevance of lung ultrasound in the diagnosis of acute respiratory failure: the BLUE protocol. Chest. 2008 Jul;134(1):117-25. doi: 10.1378/chest.07-2800. Epub 2008 Apr 10. PMID 18403664
- [Background] Malek R, Soufi S. Pulmonary Edema. 2023 Apr 7. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK557611/ PMID 32491543
- [Background] Singbartl K, Kellum JA. AKI in the ICU: definition, epidemiology, risk stratification, and outcomes. Kidney Int. 2012 May;81(9):819-25. doi: 10.1038/ki.2011.339. Epub 2011 Oct 5. PMID 21975865
- [Background] Kobbe P, Vodovotz Y, Kaczorowski DJ, Billiar TR, Pape HC. The role of fracture-associated soft tissue injury in the induction of systemic inflammation and remote organ dysfunction after bilateral femur fracture. J Orthop Trauma. 2008 Jul;22(6):385-90. doi: 10.1097/BOT.0b013e318175dd88. PMID 18594302
- [Background] Sikka G, Miller KL, Steppan J, Pandey D, Jung SM, Fraser CD 3rd, Ellis C, Ross D, Vandegaer K, Bedja D, Gabrielson K, Walston JD, Berkowitz DE, Barouch LA. Interleukin 10 knockout frail mice develop cardiac and vascular dysfunction with increased age. Exp Gerontol. 2013 Feb;48(2):128-35. doi: 10.1016/j.exger.2012.11.001. Epub 2012 Nov 13. PMID 23159957
- [Background] Vadivelu N, Chang D, Helander EM, Bordelon GJ, Kai A, Kaye AD, Hsu D, Bang D, Julka I. Ketorolac, Oxymorphone, Tapentadol, and Tramadol: A Comprehensive Review. Anesthesiol Clin. 2017 Jun;35(2):e1-e20. doi: 10.1016/j.anclin.2017.01.001. Epub 2017 Apr 14. PMID 28526155
- [Background] Rogero MM, Calder PC. Obesity, Inflammation, Toll-Like Receptor 4 and Fatty Acids. Nutrients. 2018 Mar 30;10(4):432. doi: 10.3390/nu10040432. PMID 29601492
- [Background] Almahmoud K, Namas RA, Abdul-Malak O, Zaaqoq AM, Zamora R, Zuckerbraun BS, Sperry J, Peitzman AB, Billiar TR, Vodovotz Y. Impact of Injury Severity on Dynamic Inflammation Networks Following Blunt Trauma. Shock. 2015 Aug;44(2):101-9. doi: 10.1097/SHK.0000000000000395. PMID 26009819
- [Background] Namas RA, Vodovotz Y, Almahmoud K, Abdul-Malak O, Zaaqoq A, Namas R, Mi Q, Barclay D, Zuckerbraun B, Peitzman AB, Sperry J, Billiar TR. Temporal Patterns of Circulating Inflammation Biomarker Networks Differentiate Susceptibility to Nosocomial Infection Following Blunt Trauma in Humans. Ann Surg. 2016 Jan;263(1):191-8. doi: 10.1097/SLA.0000000000001001. PMID 25371118
- [Background] Xiao W, Mindrinos MN, Seok J, Cuschieri J, Cuenca AG, Gao H, Hayden DL, Hennessy L, Moore EE, Minei JP, Bankey PE, Johnson JL, Sperry J, Nathens AB, Billiar TR, West MA, Brownstein BH, Mason PH, Baker HV, Finnerty CC, Jeschke MG, Lopez MC, Klein MB, Gamelli RL, Gibran NS, Arnoldo B, Xu W, Zhang Y, Calvano SE, McDonald-Smith GP, Schoenfeld DA, Storey JD, Cobb JP, Warren HS, Moldawer LL, Herndon DN, Lowry SF, Maier RV, Davis RW, Tompkins RG; Inflammation and Host Response to Injury Large-Scale Collaborative Research Program. A genomic storm in critically injured humans. J Exp Med. 2011 Dec 19;208(13):2581-90. doi: 10.1084/jem.20111354. Epub 2011 Nov 21. PMID 22110166
- [Background] Pape HC, Marcucio R, Humphrey C, Colnot C, Knobe M, Harvey EJ. Trauma-induced inflammation and fracture healing. J Orthop Trauma. 2010 Sep;24(9):522-5. doi: 10.1097/BOT.0b013e3181ed1361. PMID 20736786
- [Background] Mazzocca AD, McCarthy MB, Intravia J, Beitzel K, Apostolakos J, Cote MP, Bradley J, Arciero RA. An in vitro evaluation of the anti-inflammatory effects of platelet-rich plasma, ketorolac, and methylprednisolone. Arthroscopy. 2013 Apr;29(4):675-83. doi: 10.1016/j.arthro.2012.12.005. Epub 2013 Feb 6. PMID 23395471
- [Background] Zhang W, Mei R, Wu S. Ketorolac tromethamine represses senescence in aging articular chondrocytes. Biosci Biotechnol Biochem. 2022 Jun 25;86(7):837-845. doi: 10.1093/bbb/zbac047. PMID 35404445
- [Background] Carvalho B, Lemmens HJ, Ting V, Angst MS. Postoperative subcutaneous instillation of low-dose ketorolac but not hydromorphone reduces wound exudate concentrations of interleukin-6 and interleukin-10 and improves analgesia following cesarean delivery. J Pain. 2013 Jan;14(1):48-56. doi: 10.1016/j.jpain.2012.10.002. Epub 2012 Dec 4. PMID 23218935
- [Background] Kim MH, Hahm TS. Plasma levels of interleukin-6 and interleukin-10 are affected by ketorolac as an adjunct to patient-controlled morphine after abdominal hysterectomy. Clin J Pain. 2001 Mar;17(1):72-7. doi: 10.1097/00002508-200103000-00010. PMID 11289091
- [Background] Singh P, Rastogi S, Bansal M, Kumar S, Singh R, Nishad SG, Reddy MP, Anand KR, Kumar S, Thayath MN. A prospective study to assess the levels of interleukin-6 following administration of diclofenac, ketorolac and tramadol after surgical removal of lower third molars. J Maxillofac Oral Surg. 2015 Jun;14(2):219-25. doi: 10.1007/s12663-013-0609-1. Epub 2014 Feb 18. PMID 26028838
- [Background] Kuchalik J, Magnuson A, Tina E, Gupta A. Does local infiltration analgesia reduce peri-operative inflammation following total hip arthroplasty? A randomized, double-blind study. BMC Anesthesiol. 2017 May 3;17(1):63. doi: 10.1186/s12871-017-0354-y. PMID 28468607
- [Background] Namas RA, Almahmoud K, Mi Q, Ghuma A, Namas R, Zaaqoq A, Zhu X, Abdul-Malak O, Sperry J, Zamora R, Billiar TR, Vodovotz Y. Individual-specific principal component analysis of circulating inflammatory mediators predicts early organ dysfunction in trauma patients. J Crit Care. 2016 Dec;36:146-153. doi: 10.1016/j.jcrc.2016.07.002. Epub 2016 Jul 11. PMID 27546764
- [Background] Levy RM, Mollen KP, Prince JM, Kaczorowski DJ, Vallabhaneni R, Liu S, Tracey KJ, Lotze MT, Hackam DJ, Fink MP, Vodovotz Y, Billiar TR. Systemic inflammation and remote organ injury following trauma require HMGB1. Am J Physiol Regul Integr Comp Physiol. 2007 Oct;293(4):R1538-44. doi: 10.1152/ajpregu.00272.2007. Epub 2007 Jul 25. PMID 17652366
- [Background] Giannoudis PV, Giannoudi M, Stavlas P. Damage control orthopaedics: lessons learned. Injury. 2009 Nov;40 Suppl 4:S47-52. doi: 10.1016/j.injury.2009.10.036. PMID 19895952
- [Background] Billiar TR, Hunt BJ, Bailly S. Targeting inflammation in traumatic injury: entering a new era. Intensive Care Med. 2023 Aug;49(8):977-978. doi: 10.1007/s00134-023-07152-2. Epub 2023 Jul 19. No abstract available. PMID 37466669
- [Background] Namas R, Ghuma A, Hermus L, Zamora R, Okonkwo DO, Billiar TR, Vodovotz Y. The acute inflammatory response in trauma / hemorrhage and traumatic brain injury: current state and emerging prospects. Libyan J Med. 2009 Sep 1;4(3):97-103. doi: 10.4176/090325. PMID 21483522
- [Background] Giannoudis PV, Hak D, Sanders D, Donohoe E, Tosounidis T, Bahney C. Inflammation, Bone Healing, and Anti-Inflammatory Drugs: An Update. J Orthop Trauma. 2015 Dec;29 Suppl 12:S6-9. doi: 10.1097/BOT.0000000000000465. PMID 26584270
- [Background] Dodwell ER, Latorre JG, Parisini E, Zwettler E, Chandra D, Mulpuri K, Snyder B. NSAID exposure and risk of nonunion: a meta-analysis of case-control and cohort studies. Calcif Tissue Int. 2010 Sep;87(3):193-202. doi: 10.1007/s00223-010-9379-7. Epub 2010 Jun 15. PMID 20552333
- [Result] Foster JA, Kavolus MW, Landy DC, Pectol RW, Sneed CR, Kinchelow DL, Griffin JT, Hawk GS, Bernard AC, Oyler DR, Aneja A. Low-Dose Short-Term Scheduled Ketorolac Reduces Opioid Use and Pain in Orthopaedic Polytrauma Patients: A Randomized Clinical Trial. J Orthop Trauma. 2023 Dec 1;37(12):633-639. doi: 10.1097/BOT.0000000000002703. PMID 37752630
- [Result] Foster JA, Hawk GS, Landy DC, Griffin JT, Bernard AC, Oyler DR, Southall WGS, Muhammad M, Sierra-Arce CR, Mounce SD, Borgida JS, Xiang L, Aneja A. Does Scheduled Low-Dose Short-Term NSAID (Ketorolac) Modulate Cytokine Levels After Orthopaedic Polytrauma? A Secondary Analysis of a Randomized Clinical Trial. J Orthop Trauma. 2024 Jul 1;38(7):358-365. doi: 10.1097/BOT.0000000000002807. PMID 38506517
- See also: Pilot Study Results #1 — https://journals.lww.com/jorthotrauma/fulltext/2023/12000/low_dose_short_term_scheduled_ketorolac_reduces.7.aspx
- See also: Pilot Study Results #2 — https://journals.lww.com/jorthotrauma/abstract/9900/does_scheduled_low_dose_short_term_nsaid.357.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After obtaining institutional review board approval at a single Level I trauma center and clinical trial registration (ClinicalTrials.gov; NCT03671746), potential subjects were screened, recruited, and enrolled from February 2019 to October 2022. The types of locations in which participants were enrolled included the institution's emergency department, pre-operative holding area, or hospital unit.
Pre-assignment Details: No enrolled participants were excluded from the study before assignment to groups.
Groups:
- Standard of Care With NSAID: Participants in the group will receive Ketorolac in addition to standard of care for the standard Advanced Trauma Life Support (ATLS) or ICU routine medical care.
  Ketorolac: Participants will receive Ketorolac at 15 mg IV every 6 hours for their first 5 days of hospitalization
Period: Overall Study
Arm/Group | Standard of Care Without NSAID | Standard of Care With NSAID
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care Without NSAID: Polytrauma participants will receive standard of care in addition to saline solution according to standard ATLS and standard ICU routine medical care.
  Saline Solution: Participants will receive 1 ml of saline solution IV every 6 hours for their first 5 days of hospitalization
- Standard of Care With NSAID: Participants in the group will receive Ketorolac in addition to standard of care for the standard ATLS or ICU routine medical care.
  Ketorolac: Participants will receive Ketorolac at 15 mg IV every 6 hours for their first 5 days of hospitalization
- Total: Total of all reporting groups
Arm/Group | Standard of Care Without NSAID | Standard of Care With NSAID | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (16.2) | 39.5 (17.2) | 39.8 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 24 | 21 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 35 | 35 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 33 | 33 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.5 (6.4) | 28.2 (7.3) | 28.9 (6.8)
New Injury Severity Score (NISS) [Mean (Standard Deviation); unit: units on a scale] — The New Injury Severity Score (NISS) is a modification of the Injury Severity Score (ISS), which serves as a scale for determining injury burden in polytrauma patients. To calculate the NISS, the sum of squares of the three most severe injuries are calculated, regardless of body region. Each injury is scored from 0 to 3, with 3 being the most severe. Since the sum of squares of the three most severe injuries is calculated, this provides a NISS scale of 0 to 27, with 0 being no injury to 27 being the most severe injury burden.
  units on a scale | 15.1 (6.4) | 14.0 (5.2) | 14.6 (5.8)
Surgery Count [Mean (Standard Deviation); unit: number of surgeries] | 1.4 (0.7) | 1.2 (0.6) | 1.3 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospital Stay
Description: Duration of the hospital stay will be calculated from electronic health record
Time Frame: Up to 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard of Care Without NSAID | Standard of Care With NSAID
Number analyzed (Participants) | 35 | 35
days | 7 [3 to 10] | 8 [4.5 to 11.5]
Statistical Analysis 1: Comparison: Standard of Care Without NSAID vs Standard of Care With NSAID; Sample size calculations were performed using Length of Stay (LOS) as this was the primary outcome. Using a significance level of 0.05 and assumed standard deviation of 1.5 days, a sample size of 42 patients/group (84 total) would yield 80% power to detect a difference of 0.928 days in average LOS between groups. Allowing for a dropout rate of up to 25%, recruitment was planned for 56 patients/group. Power calculations were performed using nQuery 8.5 (Statistical Solutions Ltd; Cork, Ireland); Test type: Superiority; p = 0.275, ANOVA; A Kenward-Roger adjustment was used to correct for negative bias in the standard errors and degrees of freedom calculations; Median Difference (Final Values) = 1.5, Standard Deviation 1.5

2. Secondary Outcome: Morphine Milligram Equivalents in House
Description: The the morphine milligram equivalents (MME) will be recorded throughout the course of the hospital stay. These will be reported as daily totals.
Time Frame: Hospital Day 0 (Enrollment), Day 1, Day 2, Day 3, Day 4, Day 5
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalents
Arm/Group | Standard of Care Without NSAID | Standard of Care With NSAID
Number analyzed (Participants) | 35 | 35
morphine milligram equivalents
  Day 0 (Enrollment) | 82.5 [49 to 118] | 86 [38 to 120]
  Day 1 | 67.75 [48 to 81] | 48.75 [19 to 82]
  Day 2 | 62 [38 to 90] | 53 [26 to 75]
  Day 3 | 72 [45 to 99] | 38.25 [28 to 75]
  Day 4 | 60 [28 to 78] | 30 [23 to 60]
  Day 5 | 63.75 [32 to 88] | 30 [18 to 52]
Statistical Analysis 1: Comparison: Standard of Care Without NSAID vs Standard of Care With NSAID; Sample size calculations were performed using LOS as this was the primary outcome. Using a significance level of 0.05 and an assumed standard deviation of 1.5 days, a sample size of 42 patients/group (84 total) would yield 80% power to detect a difference of 0.928 days in average LOS between groups. Allowing for a dropout rate of up to 25%, recruitment was originally planned for 56 patients/group. Power calculations were performed using nQuery 8.5 (Statistical Solutions Ltd; Cork, Ireland); Test type: Superiority; p < 0.05, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Change in Patient Pain Scores
Description: The patient reported pain scores (visual analogue pain scores) will be recorded throughout the course of the hospital stay. The scores are reported by the patients and range from 0 indicating no pain to 100 meaning the worst pain imaginable. These will be reported as daily averages.
Time Frame: Hospital Day 0 (Enrollment), Day 1, Day 2, Day 3, Day 4, Day 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care Without NSAID | Standard of Care With NSAID
Number analyzed (Participants) | 35 | 35
score on a scale
  Day 0 (Enrollment) | 55.1 (27.5) | 68.2 (24.4)
  Day 1 | 52.2 (31.3) | 42.7 (25.6)
  Day 2 | 53.9 (26.5) | 47.4 (27.7)
  Day 3 | 54.1 (27.3) | 56.3 (26.0)
  Day 4 | 59.5 (26.9) | 43.3 (24.0)
  Day 5 | 59.2 (25.6) | 52.6 (21.9)
Statistical Analysis 1: Comparison: Standard of Care Without NSAID vs Standard of Care With NSAID; Sample size calculations were performed regarding LOS as this was the primary outcome measure. Using a significance level of 0.05 and an assumed SD of 1.5 days, a sample size of 42 patients per group (84 total) would yield 80% power to detect a difference of 0.928 days in average LOS between groups. Allowing for a dropout rate of up to 25%, recruitment was originally planned for 56 patients per group. Power calculations were performed using nQuery 8.5 (Statistical Solutions Ltd; Cork, Ireland); Test type: Superiority; p < 0.05, Mixed Models Analysis; The VAS model was adjusted for baseline levels as a covariate, which differed significantly between groups

4. Secondary Outcome: Change in Interleukin 1a
Description: Daily blood collections during the first 5 days of hospitalization. Interleukin 1a will be measured by the sandwich ELISA, and data will be presented as change in the baseline level of Interleukin 1 from presentation to the emergency room to day 5 of hospitalization.
Time Frame: Hospital Day 0 (Enrollment), Day 1, Day 2, Day 3, Day 4, Day 5
Population: The cytokine analysis was limited to only short-term inpatient data collected from the date of admission to inpatient Day 3. While research personnel attempted to recruit patients with anticipated hospital stays of at least five days, there was a notable decrease in hospitalized subjects past Day 3. To maintain study power and make meaningful conclusions, the authors decided to present findings analyzed during the first three hospital days.
Measure: Median (Inter-Quartile Range); unit: fg/mL
Arm/Group | Standard of Care Without NSAID | Standard of Care With NSAID
Number analyzed (Participants) | 33 | 31
fg/mL
  Day 0 (Enrollment) | 115.1 [82 to 164] | 138.8 [65 to 177]
  Day 1 | 112.7 [72 to 176] | 122.6 [79 to 169]
  Day 2 | 119.3 [78 to 179] | 135.4 [60 to 207]
  Day 3 | 104.2 [76 to 153] | 135.0 [45 to 189]
  Day 4: number analyzed (Participants) | 16 | 17
  Day 4 | 150.2 [74 to 180] | 85.2 [23 to 203]
  Day 5: number analyzed (Participants) | 13 | 16
  Day 5 | 101.9 [65 to 162] | 148.7 [77 to 176]
Statistical Analysis 1: Comparison: Standard of Care Without NSAID vs Standard of Care With NSAID; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.564, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Group-level summary statistics were calculated for demographic and clinical variables, and differences between groups were evaluated using two-sample t-tests for quantitative measures and Fisher's exact tests for categorical measures, as appropriate. Time and group comparisons for each cytokine were made using linear mixed models, with and without adjusting for selected covariates. Patient demographic variables and clinical outcomes of interest were considered for inclusion as covariates in each model but were only retained if they significantly improved the model. Linear mixed models were log-transformed, double-log-transformed, or square-root-transformed to correct for right skewness, as appropriate. Likelihood ratio testing and Akaike information criterion were used to select appropriate covariance structures in each case. All analyses were completed in SAS 9.4 (SAS Institute Inc.; Cary, NC, USA)

5. Secondary Outcome: Change in Interleukin 1b
Description: Daily blood collections during the first 5 days of hospitalization. Interleukin 1b will be measured by the sandwich ELISA, and data will be presented as change in the baseline level of Interleukin 1 from presentation to the emergency room to day 5 of hospitalization.
Time Frame: Hospital Day 0 (Enrollment), Day 1, Day 2, Day 3, Day 4, Day 5
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Standard of Care Without NSAID | Standard of Care With NSAID
Number analyzed (Participants) | 32 | 32
pg/mL
  Day 0 (Enrollment) | 0.119 [0.073 to 0.165] | 0.119 [0.085 to 0.187]
  Day 1 | 0.095 [0.043 to 0.184] | 0.130 [0.070 to 0.199]
  Day 2 | 0.084 [0.058 to 0.132] | 0.118 [0.080 to 0.230]
  Day 3 | 0.091 [0.068 to 0.141] | 0.108 [0.072 to 0.276]
  Day 4: number analyzed (Participants) | 16 | 17
  Day 4 | 0.064 [0.048 to 0.097] | 0.166 [0.091 to 0.216]
  Day 5: number analyzed (Participants) | 13 | 16
  Day 5 | 0.056 [0.043 to 0.071] | 0.126 [0.081 to 0.184]
Statistical Analysis 1: Comparison: Standard of Care Without NSAID vs Standard of Care With NSAID; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.118, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; [other analysis details as in outcome 4, analysis 1]

6. Secondary Outcome: Change in Interleukin 6
Description: Daily blood collections during the first 5 days of hospitalization. Interleukin 6 will be measured by the sandwich ELISA, and data will be presented as change in the baseline level of Interleukin 6 from presentation to the emergency room to day 5 of hospitalization.
Time Frame: Hospital Day 0 (Enrollment), Day 1, Day 2, Day 3, Day 4, Day 5
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Standard of Care Without NSAID | Standard of Care With NSAID
Number analyzed (Participants) | 33 | 32
pg/mL
  Day 0 (Enrollment) | 21.5 [16 to 27] | 20.6 [13 to 25]
  Day 1 | 21.2 [10 to 38] | 14.6 [8 to 34]
  Day 2 | 16.3 [8 to 26] | 11.9 [6 to 18]
  Day 3 | 12.9 [6 to 20] | 11.2 [6 to 27]
  Day 4: number analyzed (Participants) | 16 | 17
  Day 4 | 7.9 [6 to 15] | 10.5 [7 to 23]
  Day 5: number analyzed (Participants) | 13 | 16
  Day 5 | 10.5 [8 to 20] | 10.8 [5 to 26]
Statistical Analysis 1: Comparison: Standard of Care Without NSAID vs Standard of Care With NSAID; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.215, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; [other analysis details as in outcome 4, analysis 1]

7. Secondary Outcome: Change in Interleukin 10
Description: Daily blood collections during the first 5 days of hospitalization. Interleukin 10 will be measured by the sandwich ELISA, and data will be presented as change in the baseline level of Interleukin 10 from presentation to the emergency room to day 5 of hospitalization.
Time Frame: Hospital Day 0 (Enrollment), Day 1, Day 2, Day 3, Day 4, Day 5
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Standard of Care Without NSAID | Standard of Care With NSAID
Number analyzed (Participants) | 33 | 32
pg/mL
  Day 0 (Enrollment) | 1.10 [0.7 to 1.7] | 1.11 [0.8 to 2.3]
  Day 1 | 0.90 [0.6 to 1.6] | 0.76 [0.5 to 1.1]
  Day 2 | 0.57 [0.4 to 1.3] | 0.62 [0.4 to 1.1]
  Day 3 | 0.65 [0.5 to 0.9] | 0.64 [0.5 to 1.5]
  Day 4: number analyzed (Participants) | 16 | 17
  Day 4 | 0.49 [0.4 to 0.8] | 0.59 [0.5 to 0.9]
  Day 5: number analyzed (Participants) | 13 | 16
  Day 5 | 0.72 [0.4 to 1.3] | 0.75 [0.4 to 1]
Statistical Analysis 1: Comparison: Standard of Care Without NSAID vs Standard of Care With NSAID; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.043, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; [other analysis details as in outcome 4, analysis 1]

8. Secondary Outcome: Change in Prostaglandin E-2
Description: Blood will be collected over the course of 5 days of hospitalization. Prostaglandin E-2 will be measured by the sandwich ELISA, and data will be presented as change in the baseline level of Prostaglandin E-2 from presentation to the emergency room to day 5 of hospitalization
Time Frame: Hospital Day 0 (Enrollment), Day 1, Day 2, Day 3, Day 4, Day 5
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Standard of Care Without NSAID | Standard of Care With NSAID
Number analyzed (Participants) | 26 | 28
pg/mL
  Day 0 (Enrollment) | 352.2 [161 to 673] | 448.3 [232 to 738]
  Day 1 | 477.0 [309 to 810] | 375.8 [292 to 587]
  Day 2 | 345.8 [178 to 563] | 356.6 [209 to 509]
  Day 3 | 319.8 [239 to 605] | 371.3 [251 to 515]
  Day 4: number analyzed (Participants) | 13 | 13
  Day 4 | 347.6 [189 to 379] | 304.7 [237 to 430]
  Day 5: number analyzed (Participants) | 13 | 10
  Day 5 | 266.9 [209 to 475] | 322.3 [183 to 540]
Statistical Analysis 1: Comparison: Standard of Care Without NSAID vs Standard of Care With NSAID; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.617, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; [other analysis details as in outcome 4, analysis 1]

9. Secondary Outcome: Post Traumatic Complications
Description: The Incidence of post-traumatic complications in the patients which includes, but is not limited to the occurrence of pulmonary complications (i.e., bacterial pneumonia, pulmonary edema, acute respiratory failure) and AKI will be recorded throughout the duration of the hospital stay, usually up to 30 days. Data will be presented as the percentage of participants with a diagnosed post-traumatic complication.
Time Frame: Up to 30 days
Population: Two participants were excluded from the secondary analysis, as blood samples were not able to be collected from these patients. Due to a transition in our institution's electronic medical record, one patient's chart could not be recovered, hence secondary clinical outcomes could not be collected for this patient (n=67).
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Without NSAID | Standard of Care With NSAID
Number analyzed (Participants) | 33 | 34
Participants
  Pulmonary Complications | 4 | 3
  Acute Kidney Injury (AKI) | 2 | 0

10. Secondary Outcome: Mortality
Description: The Incidence of death related to the initial trauma/traumatic complications will be recorded for the first 30 days.
Time Frame: Up to 30 days
Population: Two participants were excluded from the secondary analysis, as blood samples were not able to be collected from these patients (n=68). Due to a transition in our institution's electronic medical record, one patient's chart could not be recovered, hence secondary clinical outcomes could not be collected for this patient.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Without NSAID | Standard of Care With NSAID
Number analyzed (Participants) | 33 | 34
Participants | 0 | 0
Statistical Analysis 1: Comparison: Standard of Care Without NSAID vs Standard of Care With NSAID; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.05, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; [other analysis details as in outcome 4, analysis 1]

11. Secondary Outcome: Change in Inpatient Subjective Pain Reports
Description: as for outcome 3
Time Frame: Hospital Day 0 (Enrollment), Day 1, Day 2, Day 3, Day 4, Day 5
Population: Change in patient pain scores during the hospital stay was inadvertently entered twice (as outcomes #3: Change in Patient Pain Scores and #11: Change in Inpatient Subjective Pain Reports). These represent identical outcomes which was change in patient pain during the hospital stay. Please refer to outcome #3 for the corresponding data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care Without NSAID | Standard of Care With NSAID
Number analyzed (Participants) | 35 | 35
score on a scale
  Day 0 (Enrollment) | 55.1 (27.5) | 68.2 (24.4)
  Day 1 | 52.2 (31.3) | 42.7 (25.6)
  Day 2 | 53.9 (26.5) | 47.4 (27.7)
  Day 3 | 54.1 (27.3) | 56.3 (26.0)
  Day 4 | 59.5 (26.9) | 43.3 (24.0)
  Day 5 | 59.2 (25.6) | 52.6 (21.9)

12. Secondary Outcome: Change in Outpatient Subjective Pain Reports
Description: Patient reports of level of pain and how much it inhibits their daily activities will be recorded in the outpatient setting. The scores are reported by the patients (visual analogue scale) and range from 0 indicating no pain to 100 meaning the worst pain imaginable. This will be reported for each patient follow-up visit. Several visits are possible and data will only be collected for the first year of follow-up. Data presented as the change in subject pain from baseline to 365 days.
Time Frame: up to 365 days
Population: Only nine patients completed the required follow-up, resulting in insufficient data to conduct meaningful statistical analysis or draw clinically relevant conclusions.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Standard of Care Without NSAID | Standard of Care With NSAID
Number analyzed (Participants) | 3 | 6
units on a scale | -22.7 [-40 to -1] | -16.7 [-60 to -12]

ADVERSE EVENTS:
Time Frame: Up to 30 days
Arm/Group | Standard of Care Without NSAID | Standard of Care With NSAID
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 6/35 | 3/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care Without NSAID (N=35) | Standard of Care With NSAID (N=35)
Pulmonary Complications (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) — Pulmonary complications were defined as bacterial pneumonia, pulmonary edema, or acute respiratory failure.
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 0 (0) — Acute kidney injury was defined as an increase in serum creatinine greater than or equal to 0.3 mg/dL within a 48-hour period.

LIMITATIONS AND CAVEATS:
The study was unable to achieve the target enrollment of 56 patients per group due to the institution suspending all clinical trial enrollment during the COVID-19 pandemic. Blood samples were not able to be collected from two patients and clinical outcomes for one patient. Due to a transition in the institution's electronic medical record that occurred in 2021, one patient's chart could not be recovered, hence clinical outcomes could not be collected for this patient.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-22): https://cdn.clinicaltrials.gov/large-docs/46/NCT03671746/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/46/NCT03671746/ICF_001.pdf